CLINICAL TRIAL: NCT00264641
Title: The Impact of Renin-angiotensin System on Brain Activation During Hypoglycaemia in Healthy Men, a PET Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hypoglycaemia Research Group (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Birger Thorsteinsson, Professor, Hypoglycaemia Research Group
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2005-2-15
Record Dates: First submitted 2005-12-12; First posted 2005-12-13 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Hypoglycemia; Cognitive Impairment
Keywords: Hypoglycemia; Cognitive impairment; PET; CalCAP
MeSH Terms: conditions — Hypoglycemia; Cognitive Dysfunction | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High RAS activity (Experimental): 10 healthy men were characterized by having high basal RAS activity.
  Interventions: Drug: Human insulin
- Low RAS activity (Experimental): 10 healthy men were characterized by having either a low basal RAS activity.
  Interventions: Drug: Human insulin

INTERVENTIONS:
Drug: Human insulin — Hyperinsulinaemic induced hypoglycaemia

SUMMARY:
The purpose of this study is to evaluate the cerebral blood flow in subjects with high and low activity in the renin-angiotensin system (RAS).The renin-angiotensin system is a hormone system which is involved in the regulation of the blood pressure. Earlier studies have shown that high RAS activity is associated with a more pronounced cognitive impairment during hypoglycaemia compared to low RAS activity in both type 1 diabetic patients and healthy volunteers. We intend to examine brain activity by oxygen-15 labelled water-PET scanning during hypoglycaemia in response to cognitive function testing in 20 healthy male volunteers with high and low RAS activity, respectively

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the regional cerebral blood flow in subjects with high and low activity in the renin-angiotensin system (RAS). Earlier studies have shown that high RAS activity is associated with a more pronounced cognitive impairment during hypoglycaemia compared to low RAS activity in both type 1 diabetic patients and healthy volunteers. We intend to examine brain activity by oxygen-15 labelled water-PET scanning during hypoglycaemia in response to cognitive function testing in 20 healthy male volunteers with high and low RAS activity, respectively.

ELIGIBILITY:
Inclusion Criteria:Male Age 18-40 years Right-handed In good general health based on history High/low RAS activity (high ACE activity, A-allele for angiotensin II receptor (subtype 2) and high plasma angiotensinogen, or low ACE activity, low plasma angiotensinogen and not carrier of the A-allele for angiotensin II receptor (subtype 2)).

-

Exclusion Criteria:

Any evidence of mental, neurological or medical illnesses. The presence of ferromagnetic metal in the body. Claustrophobia Exposure to radiation within the last year

-

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2006-01; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Birger Thorsteinsson, MD, DMSci, Study Chair — Hypoglycaemia Research Group
Locations (1):
- Medical Department I, Hillerød Hospital, Hillerød, Hillerød, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bie-Olsen LG, Pedersen-Bjergaard U, Kjaer TW, Lonsdale MN, Law I, Thorsteinsson B. Association between regional cerebral blood flow during hypoglycemia and genetic and phenotypic traits of the renin-angiotensin system. J Cereb Blood Flow Metab. 2009 Nov;29(11):1790-5. doi: 10.1038/jcbfm.2009.94. Epub 2009 Jul 8. PMID 19584889
- [Result] Bie-Olsen LG, Pedersen-Bjergaard U, Kjaer TW, Lonsdale MN, Law I, Thorsteinsson B. Differences in cortical and pituitary activity in response to hypoglycaemia and cognitive testing in healthy men with different basal activity of the renin-angiotensin system. J Renin Angiotensin Aldosterone Syst. 2010 Sep;11(3):173-9. doi: 10.1177/1470320310364182. Epub 2010 Mar 9. PMID 20215476
- [Result] Bie-Olsen LG, Kjaer TW, Pedersen-Bjergaard U, Lonsdale MN, Holst JJ, Law I, Thorsteinsson B. Changes of cognition and regional cerebral activity during acute hypoglycemia in normal subjects: A H2 15O positron emission tomographic study. J Neurosci Res. 2009 Jun;87(8):1922-8. doi: 10.1002/jnr.22002. PMID 19170163

RESULTS

PARTICIPANT FLOW:
Groups:
- High RAS Activity: High RAS was defined as serum ACE and plasma angiotensinogen concentration in the highest quartiles in the population combined with AT2 receptor genotype A
- Low RAS Activity: Low RAS was defined as serum ACE and plasma angiotensinogen concentration in the lowest quartiles in the population combined with AT2 receptor genotype G
Period: Overall Study
Arm/Group | High RAS Activity | Low RAS Activity
Started | 10 | 10
Initiation of the Study | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- High RAS Activity: High RAS activity is defined in the protocol
- Low RAS Activity: Low RAS activity is defined in the protocol
- Total: Total of all reporting groups
Arm/Group | High RAS Activity | Low RAS Activity | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (4.8) | 27 (5.6) | 26.5 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Only men were included
  Participants
    Female | 0 | 0 | 0
    Male | 10 | 10 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Denmark | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Cerebral Activation During Hypoglycaemia
Description: To compare the high RAS activity vs low RAS activity a Z score was used.
Time Frame: After 4 scans on day 1
Population: Only data available is between group analysis
Measure: Number; unit: Z score
Groups:
- All Study Participants: From a screening population ten subjects with high RAS activity - defined as serum ACE and plasma angiotensinogen concentrations in the highest quartile in the population combined with presence of AT2 receptor genotype A corresponding to low expression of the receptor (maximum stimulation via the AT1 receptor) - were selected And 10 males with low RAS activity - defined as serum ACE and plasma angiotensinogen concentrations in the lowest quartile in the population combined with the presence of AT2 receptor genotype G corresponding to high expression of the receptor (58) (minimum stimulation via the AT1 receptor) were selected
Arm/Group | All Study Participants
Number analyzed (Participants) | 20
Z score
  Low RAS>High RAS Right sup frontal gyrus | 4.85
  High RAS>Low RAS post entorhinal cortex | 4.55

ADVERSE EVENTS:
Groups:
- High RAS Activity: High RAS activity is described in the protocol
- Low RAS Activity: Low RAS activity is described in the protocol
Arm/Group | High RAS Activity | Low RAS Activity
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes